CLINICAL TRIAL: NCT04320706
Title: Oral Oxytocin Modulation of Brain and Behavioral Responses to Emotional Stimuli in Healthy Men
Brief Title: Oral Oxytocin Modulation of Responses to Emotional Stimuli
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Principal Investigator, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-60
Record Dates: First submitted 2020-03-21; First posted 2020-03-25 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Healthy
Keywords: oral Oxytocin; emotional processing; anxiety; reward
MeSH Terms: conditions — Anxiety Disorders | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind between-subject design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Oxytocin (Experimental): Oxytocin orally (24 IU)
  Interventions: Drug: Oral Oxytocin
- Oral Placebo (Placebo Comparator): Placebo orally (identical ingredients, except the active agent)
  Interventions: Drug: Oral Placebo

INTERVENTIONS:
Drug: Oral Oxytocin — Administration of oxytocin (24 international units) orally
  Arms: Oral Oxytocin
Drug: Oral Placebo — Administration of placebo orally
  Arms: Oral Placebo

SUMMARY:
The main aim of the study is to investigate whether orally administered oxytocin (24IU) can modulate neural and behavioral responses to positive and negative valence stimuli during basal (emotional scenes) and higher order (facial stimuli) emotional processing.

DETAILED DESCRIPTION:
A number of previous studies have reported both neural and social cognition effects of intranasally administered oxytocin, although it is unclear whether functional effects are mediated by the peptide directly entering the brain or indirectly via raising peripheral concentrations. The investigators hypothesize that one method of producing a similar pattern of increased peripheral oxytocin concentrations but without the possibility of direct entry into the brain would be to administer the peptide lingually. In the current double-blind, between-subject, placebo controlled study 80 healthy male subjects will be recruited and receive either oxytocin (24IU) or placebo control administered orally (lingual). 45 minutes after treatment subjects will be required to complete both face emotion and emotional scene processing tasks during fMRI scanning. After the tasks, subjects will be required to rate their valence, intensity and arousal response to the same emotional face and scene stimuli which were presented during MRI acquisition. Blood samples will be taken before and 30 min after the oral treatment interventions to assess oxytocin blood concentrations. All subjects will be asked to complete a range of questionnaires before treatment to control for possible pre-treatment confounders in terms of personality traits and mood: Beck Depression Inventory II (BDI), Autism Spectrum Quotient (ASQ), Liebowitz Social Anxiety Scale (LSAS), State-Trait Anxiety Inventory (STAI), Childhood Trauma Questionnaire (CTQ), the Second Version of Social Responsiveness Scale(SRS-2), and Interpersonal Reactivity Index (IRI).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any past or present psychiatric or neurological disorders

Exclusion Criteria:

* History of brain injury
* Head trauma
* Substance abuse
* Medication
* fMRI contraindications (e.g. metal implants)

Ages: 17 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Effect of oral oxytocin administration of oxytocin on neural responses to positive and negative valence emotional faces, as assessed by task fMRI | 45-90 minutes after treatment
  Comparison of neural activation as assessed by functional MRI on the whole brain level between oral administration of oxytocin and placebo by means of treatment (oxytocin, placebo) x emotion (happy, neutral, angry, fear) ANOVAs and emotion-specific comparisons between the treatment groups. We hypothesized that if the effects of oxytocin administration reported following intranasal administration are primarily produced via an increase in peripheral concentrations then oral administration should produce similar effects on neural systems involved in emotional and brain reward processing. If on the other hand some, or all, of the effects of intranasal oxytocin are mediated via a direct action on the brain then oral administration should result in either no effect or alternatively a different pattern of functional effects.
Effect of oral oxytocin administration on neural responses to positive and negative valence scenes, as assessed by fMRI | 45-90 minutes after treatment
  Comparison of neural activation as assessed by functional MRI on whole brain level between oral administration of oxytocin and placebo by means of treatment (oxytocin, placebo) x emotion (neutral, positive, negative) ANOVAs and emotion-specific post hoc comparisons between the treatment groups. We hypothesize that if the effects of oxytocin administration reported following intranasal administration are primarily produced via an increase in peripheral concentrations then oral administration should produce similar effects on neural systems involved in emotional and brain reward processing. If on the other hand some, or all, of the effects of intranasal oxytocin are mediated via a direct action on the brain then oral administration should result in either no effect or alternatively a different pattern of functional effects.
Effect of oral oxytocin administration on behavioral ratings of face emotion and scene stimuli | 45-115 minutes after treatment
  Comparison of behavioral ratings of valence, arousal and intensity (9-point Likert scale) for emotional face and social scene stimuli presented again post-scan will be performed in oxytocin versus placebo control groups. We hypothesize that if the effects of oxytocin administration reported following intranasal administration are primarily produced via an increase in peripheral concentrations then oral administration should produce similar effects on behavioral ratings of positive and negative valence emotional stimuli. If on the other hand some, or all, of the effects of intranasal oxytocin are mediated via a direct action on the brain then oral administration should result in either no effect or alternatively in a different pattern of functional effects.
Change in blood oxytocin concentrations following oral administration of oxytocin | 30 minutes before treatment and 30 minutes after treatment
  Changes in blood concentrations of oxytocin from baseline after oral oxytocin treatment will be assessed by comparison with the placebo group. We hypothesize that oral oxytocin should produce a significant increase in blood oxytocin concentrations after 30 minutes.

SECONDARY OUTCOMES:
Correlations between neural responses/functional connectivity changes and post-scan behavioral ratings | 45-115 minutes after treatment
  Correlations between neural responses changes and post-scan behavioral ratings of positive and negative valence stimuli will be performed using Pearson correlation in both oxytocin and placebo groups. We hypothesize that neural responses and behavioral ratings will be correlated.
Correlations between neural responses/functional connectivity in response to positive and negative valence stimuli and basal and oral administration evoked changes in blood concentrations of oxytocin | 30 minutes before treatment to 90 minutes after treatment
  Correlations between neural responses in response to positive and negative valence stimuli and basal and oral administration evoked changes in blood concentrations of oxytocin will be performed using Pearson correlation in both oxytocin and placebo groups. We hypothesize that neural responses to emotional stimuli will correlate with basal and/or oral administration evoked oxytocin concentrations.
Correlations between behavioral ratings of positive and negative valence stimuli and basal and oral administration evoked changes in blood oxytocin concentrations | 30 minutes before treatment to 115 minutes after treatment
  Correlations between behavioral ratings of positive and negative valence stimuli and basal and oral administration evoked changes in blood oxytocin concentrations will be performed using Pearson correlation in both oxytocin and placebo groups. We hypothesize that behavioral ratings to emotional stimuli will correlate with basal and/or oral administration evoked oxytocin concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, PhD, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- school of life science and technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China